CLINICAL TRIAL: NCT01092715
Title: A Comparison of Cervical Spine Mobilization and "Standard" Physical Therapy Intervention in the Treatment of Chronic Neck Pain, A Pilot Study
Brief Title: Cervical Mobilization vs. Standard Physical Therapy for Chronic Neck Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Ralph Gay, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1423-02
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Last update posted 2010-03-25 (Estimated); Status verified 2010-03

CONDITIONS: Neck Pain
Keywords: Neck pain; Spinal manipulation; Massage
MeSH Terms: conditions — Neck Pain | interventions — Massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mobilization (Experimental): Spinal mobilization and exercises
  Interventions: Procedure: Spinal mobilization; Procedure: Neck exercises
- Massage (Active Comparator): Neck massage and exercises
  Interventions: Procedure: Massage; Procedure: Neck exercises

INTERVENTIONS:
Procedure: Spinal mobilization — Non thrust mobilization to the cervical spine
  Arms: Mobilization
Procedure: Massage — Sedative massage to cervical paraspinal muscles
  Arms: Massage
Procedure: Neck exercises — Range of motion exercises to include foraminal opening

SUMMARY:
Neck pain is a common problem in our society, accounting for 20% of all chiropractic visits. Physical therapy interventions for chronic neck pain have been chosen based on the patient's symptoms and examination findings. These interventions include superficial and deep heat, massage, traction, manual therapy, and exercise programs. There is little controlled research addressing the efficacy of these therapies. Although many of these interventions provide some patients with pain relief and increased function, studies often utilize multiple interventions on the same subject such as heat, ultrasound, cervical traction, range of motion exercises, making interpretation of the results difficult. Much of the literature to date has focused on studies of subjects suffering from acute neck pain. Many of these studies suggest that subjects report decreased pain, decreased disability and increased cervical spine active range of motion. There are no controlled studies comparing the effects of spinal mobilization and standard physical therapy on subjects with chronic neck pain. The object of this study is two fold: 1) to determine the score variability of two neck disability questionnaires )both baseline and change scores) to be used in sample size calculations, and 2) to establish the ability to recruit, treat and follow sufficient numbers of subjects needed for a full clinical trial. The ability to predict outcomes of neck pain treatment will lead to more appropriate therapies and an avoidance of unnecessary treatments.

DETAILED DESCRIPTION:
Background and Purpose: Chronic neck pain is a common problem. Studies of physical therapy for neck pain often utilize multiple interventions on the same subject making interpretation of the results difficult. The objectives of this study were two fold, 1) to establish the ability to recruit and treat subjects needed for a clinical trial of mobilization vs. massage for neck pain and 2) to estimate the variability of the Neck Disability Index (NDI) in a defined population of patients with neck pain and determine sample size for a trial. Subjects and

Methods: Subjects were randomized to either sedative massage (SM) to the neck and upper back or joint mobilization to the cervical spine (JM). All subjects also received moist heat and a home exercise program. Outcomes tracked for establishing trial feasibility included the number of referrals, number of referrals meeting inclusion criteria, number of subjects declining to participate and reasons for their refusal, acceptance rate of randomization, number of dropouts, and reasons for dropout. Descriptive statistics and baseline data were analyzed with means and standard deviations when appropriate. Groups were compared in regard to demographic and clinical characteristics only. The Neck Disability Index scores were calculated for pre-treatment, post-treatment, and change scores within each group.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain of at least 12 weeks duration

Exclusion Criteria:

* Signs and/or symptoms of cervical radiculopathy or myelopathy
* Symptomatic shoulder pathology
* History of cervical spine surgery
* History of motor vehicle collision within the past three years
* Recent neck or shoulder trauma
* Fibromyalgia or generalized pain syndrome
* History of cancer affecting the head or neck

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2003-06; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | 6 weeks
  Neck Disability Index score (patient generated score from questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Madson, PT, Principal Investigator — Mayo Clinic; Timothy J Madson, PT, Study Director — Mayo Clinic
Locations (1):
- Mayo Clinic Dept of Physical Medicine & Rehabilitation, Rochester, Minnesota, United States